CLINICAL TRIAL: NCT01741077
Title: The Effect of Folic Acid Supplementation and Pregnancy on the Folate Forms in Red Blood Cells
Status: Completed | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Brenda Hartman, Clinical Dietitian, The Hospital for Sick Children
Other Study IDs: 1000012134
Record Dates: First submitted 2012-11-27; First posted 2012-12-04 (Estimated); Last update posted 2013-12-05 (Estimated); Status verified 2013-12

CONDITIONS: Pregnancy
Keywords: pregnancy; folic acid supplementation; reproduction; folate
MeSH Terms: interventions — Folic Acid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- pregnant women: pregnant women taking 1 mg folic acid;
  Interventions: Dietary Supplement: folic acid
- non-pregnant women: non-pregnant women taking 0mg folic acid;
- non-pregnant women 2: non-pregnant women taking 1 mg folic acid
- non-pregnant women 3: non-pregnant women taking 5 mg folic acid

INTERVENTIONS:
Dietary Supplement: folic acid — subjects take multivitamin supplement containing folic acid. Women were enrolled based on whether or not they were taking supplements.
  Groups: pregnant women

SUMMARY:
The purpose of this cross-sectional study was to examine whether or not physical changes or adaptations occur in response pregnancy or to the higher intakes of folic acid from supplementation typically consumed during the reproductive period.

DETAILED DESCRIPTION:
Higher folate requirements during pregnancy to support growth and development are well established but it is unknown what metabolic changes occur in 1-carbon metabolism to provide sufficient nucleotides for DNA/RNA synthesis. Periconceptual folic acid (FA) supplementation and fortification of the food supply have been shown to reduce the risk of pregnancies with neural tube defects but conversely expose women to high FA intakes for extended periods of time. The purpose of this cross-sectional study is to establish if physiological adaptations occur in folate metabolism in response to pregnancy or higher intakes of FA typically consumed among women during the reproductive period. A convenience sample of thirty-two women (n=8/group) were recruited to compare the total concentrations and forms of folate (tetrahydrofolate [THF], 5-methylTHF, 5-formylTHF and 5, 10-methenylTHF) in red blood cells in four groups: a) pregnant women (PW, 30-36 weeks gestation) taking 1.0 mg of FA b) non-pregnant women (NPW) taking 0 mg of FA c) NPW taking 1.0 mg FA and d) NPW taking 5.0 mg FA. Blood samples were taken at a single time point and compared across groups. Total red blood cell concentrations were measured using both microbiological assay and liquid chromatography/tandem mass spectrometry (LC/MS/MS) analysis. LC/MS/MS analysis was used to determine folate form concentrations.

ELIGIBILITY:
Inclusion Criteria:

1. pregnant women-

   * between 30 to 36 weeks gestation
   * taking 1 mg folic acid in a multisupplement
2. non-pregnant women-

   * not pregnant
   * taking either 0, 1 or 5 mg folic acid in a multisupplement

Exclusion Criteria:

* Taking any medications known to interfere with folate absorption at the time of sampling (ie. Antibiotics [ can be enrolled into study if they will be off them at least two weeks prior to study commencement], methotrexate, aminopterin)
* Those with a history of any disorders or conditions that could interfere with folate absorption or metabolism from either dietary or supplement sources such as the history/presence clinically significant gastrointestinal disease (chronic diarrhea, inflammatory bowel disease, partial gastrectomy), unresolved GI symptoms(diarrhea/vomiting), steatorrhea or other conditions that interfere with absorption, distribution, metabolism or excretion of folic acid.
* Those with preexisting conditions (pre-existing maternal diabetes; insulin-dependent diabetes; previous child with neural tube disorder (NTD), cleft-lip/palate or heart defect; epilepsy and/or seizure disorders) that can increase the risk of pregnancy complicated by NTD.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: women of reproductive age
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2008-05; Primary Completion 2008-10 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Red blood cell folate concentrations - tetrahydrofolate (THF) | At the point of participation (this is a single visit, single test study)
  Bood samples were taken once at the point of participation and compared 1) pregnant women (between 30-36 weeks gestation) and non-pregnant women who were taking supplements 2) 0 mg folic acid 3) 1 mg FA, 4) and 5 mg FA. Those who were taking supplements were taking them for a minimum of 30 weeks.

SECONDARY OUTCOMES:
Red blood cell folate concentrations - 5-methyltetrahydrofolate (5-methylTHF) | At the point of participation (this is a single visit, single test study)
Red blood cell concentrations - 5-formyltetrahydrofolate (5-formylTHF) | At the point of participation (this is a single visit, single test study)
Red blood cell folate concentrations - 5,10-Methenyltetrahydrofolate (5,10-methenylTHF) | At the point of participation (this is a single visit, single test study)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah L O'Connor, PhD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Hartman BA, Fazili Z, Pfeiffer CM, O'Connor DL. Neither folic acid supplementation nor pregnancy affects the distribution of folate forms in the red blood cells of women. J Nutr. 2014 Sep;144(9):1364-9. doi: 10.3945/jn.113.189233. Epub 2014 Jul 2. PMID 24991041